CLINICAL TRIAL: NCT04530864
Title: Pre-surgical Ocular Surface Treatment With Intracanalicular Dexamethasone Insert and Effect on Intraocular Lens Measurement Accuracy - The PRECISION Study
Brief Title: Pre-Surgical Ocular Surface Treatment With Intracanalicular Dexamethasone Insert And Effect On Intraocular Lens Measurement Accuracy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prism Vision Group (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, Cynthia Matossian, Principal Investigator, Prism Vision Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEXTENZA OTX
Record Dates: First submitted 2020-07-23; First posted 2020-08-28 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Dry Eye Disease; Cataract Surgery; Ocular Surface Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- DEXTENZA Insert (Experimental): This prospective study will use a self controlled design for 35 eyes. Patients scheduled to undergo routine cataract surgery in at least one of their eyes will have their pre-surgical measurements performed, IOL calculated and surgery planned. Then they will receive insertion of an intracanalicular dexamethasone insert into the inferior punctum. At 2 weeks (+/- 2 days) post-insertion, patients will return for an identical set of measurements. The IOL will be calculated and the surgery planned based on post-insert data. The insert will be removed if present (manually or via saline irrigation). This self controlled design allows for greater control of potential confounders tied to participants' systemic and ocular health.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — All patients will receive pre-surgical ocular surface treatment with intracanalicular sustained release dexamethasone, 0.4 mg

SUMMARY:
This prospective study will use a self controlled design for 35 eyes. Patients scheduled to undergo routine cataract surgery in at least one of their eyes will have their pre-surgical measurements performed, IOL calculated and surgery planned. Then they will receive insertion of an intracanalicular dexamethasone insert into the inferior punctum. At 2 weeks (+/- 2 days) post-insertion, patients will return for an identical set of measurements. The IOL will be calculated and the surgery planned based on post-insert data. The insert will be removed if present (manually or via saline irrigation). This self controlled design allows for greater control of potential confounders tied to participants' systemic and ocular health.

DETAILED DESCRIPTION:
Ocular surface optimization is a pre-operative necessity. In cataract surgery patients, an unstable tear film reduces the quality of corneal reflections and therefore can compromise K readings, which in turn can affect the accuracy of IOL calculations and result in suboptimum refractive results. To obtain accurate measurements, patients are routinely pre-treated with a variety of medications and therapies. However, these therapies can take time, which may lead to surgical delays.

Steroids can positively impact the stability of the tear film by inhibiting and preventing ocular surface inflammation. Punctal plugs are also widely used for the treatment of dry eye manifestations, by blocking the tear drainage, increasing tear film and eye moisture. Dextenza is a sustained-release dexamethasone intracanalicular insert recently approved by the FDA for pain and inflammation post ophthalmic surgery. It is placed into the canaliculus via the lower punctum and is designed to release steroid medication for 30 days.

Previous studies have demonstrated that ocular surface disease affects the reliability of IOL calculations, potentially affecting outcomes. The insert of a punctal plug that can deliver a sustained release of dexamethasone to the eye 2 weeks (+/- 2 days) prior to final preoperative measurements may provide adequate therapy, improving the ocular surface status and, therefore, improve the reliability of IOL selection in patients undergoing cataract surgery, in a comparatively short amount of time, without introducing patient compliance barriers.

Pre-surgical measurements, IOL calculations, and surgical plans prior to the insertion of the insert will be compared to measurements, IOL calculations, and surgical plans at 2 weeks following intracanalicular dexamethasone insertion. Surgery will proceed with data from the post-insert measurements. Final refractive outcomes at one month from the second eye surgery will be compared to pre-insert data to determine refractive accuracy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Visually significant cataract
* Dry eye disease
* BCVA potential of 20/40 or better

Exclusion Criteria:

* Pregnancy
* Concurrent use of topical glaucoma medications
* Corneal scarring
* History of LASIK or PRK
* History of rigid gas permeable (RGP) lens wear
* Macular or retinal pathology requiring intervention
* Cataract surgery complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
The change in baseline data (power calculation and astigmatism management) measured by IOL Master 700 and post insert of Dextenza data (power calculation and astigmatism management) measured by IOL Master 700. | at 8 weeks (Day 0) and final refractive outcome 1 month post-op visit

SECONDARY OUTCOMES:
The change in inflammatory markers measured by MMP9 | 6 weeks BEFORE surgery from pre-insert at 8 weeks BEFORE surgery
Change in Tear Break-up Time | 6 weeks BEFORE surgery from pre-insert at 8 weeks BEFORE surgery
Change in Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED) | 6 weeks BEFORE surgery from pre-insert at 8 weeks BEFORE surgery
  The Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED) evaluates both the frequency and severity of symptoms. The patient grades the severity of her symptoms on a scale of zero to four with zero being no symptoms and four being intolerable symptoms. The numeric value for each answer is simply added with scores ranging from zero to 28. 0-4 MILD dry eye symptoms, 5-7 MODERATE dry eye symptoms, + SEVERE dry eye symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Matossian, MD, Principal Investigator — Matossian Eye Associates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epitropoulos AT, Matossian C, Berdy GJ, Malhotra RP, Potvin R. Effect of tear osmolarity on repeatability of keratometry for cataract surgery planning. J Cataract Refract Surg. 2015 Aug;41(8):1672-7. doi: 10.1016/j.jcrs.2015.01.016. PMID 26432124
- [Background] Kim P, Plugfelder S, Slomovic AR. Top 5 pearls to consider when implanting advanced-technology IOLs in patients with ocular surface disease. Int Ophthalmol Clin. 2012 Spring;52(2):51-8. doi: 10.1097/IIO.0b013e31824b4504. No abstract available. PMID 22395627
- [Background] Goldberg DF. Preoperative evaluation of patients before cataract and refractive surgery. Int Ophthalmol Clin. 2011 Spring;51(2):97-107. doi: 10.1097/IIO.0b013e31820f1f76. No abstract available. PMID 21383583
- [Background] Ale Magar JB. Comparison of the corneal curvatures obtained from three different keratometers. Nepal J Ophthalmol. 2013 Jan-Jun;5(1):9-15. doi: 10.3126/nepjoph.v5i1.7815. PMID 23584640
- [Background] Manning CA, Kloess PM. Comparison of portable automated keratometry and manual keratometry for IOL calculation. J Cataract Refract Surg. 1997 Oct;23(8):1213-6. doi: 10.1016/s0886-3350(97)80318-5. PMID 9368167